CLINICAL TRIAL: NCT04502446
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Anti-CD70 Allogeneic CRISPR-Cas9-Engineered T Cells (CTX130) in Subjects With Relapsed or Refractory T or B Cell Malignancies
Brief Title: A Safety and Efficacy Study Evaluating CTX130 in Subjects With Relapsed or Refractory T or B Cell Malignancies (COBALT-LYM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients to be followed up in the CRSP-ONC-LTF study
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-004
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: T Cell Lymphoma
Keywords: CAR T; Allogeneic; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX130 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX130

INTERVENTIONS:
Biological: CTX130 — CTX130 CD70-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components.

SUMMARY:
This is a single-arm, open-label, multicenter, Phase 1 study evaluating the safety and efficacy of CTX130 in subjects with relapsed or refractory T or B cell malignancies.

DETAILED DESCRIPTION:
The study may enroll approximately 45 subjects in total.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Age ≥18 years.
2. Confirmed diagnosis of a T cell malignancy or Diffuse Large B-Cell Lymphoma (DLBCL).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Adequate renal, liver, cardiac, and pulmonary organ function.
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX130 infusion.

Exclusion Criteria (abbreviated):

1. Prior allogeneic stem cell transplant (SCT).
2. Prior treatment with any anti-CD70 targeting agents.
3. History of certain central nervous system (CNS), cardiac or pulmonary conditions.
4. Active HIV, hepatitis B virus or hepatitis C virus infection.
5. Previous or concurrent malignancy, except treated with curative approach not requiring systemic therapy and in remission for >12 months, or any other localized malignancy with low risk of developing into metastatic disease.
6. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
7. Prior solid organ transplantation.
8. Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Part A (dose escalation) | From CTX130 infusion up to 28 days post-infusion
  Incidence of adverse events
Part B (cohort expansion) | From CTX130 infusion up to 60 months post-infusion]
  Objective response rate

SECONDARY OUTCOMES:
Progression Free Survival | From date of CTX130 infusion until date of disease progression or death due to any cause, assessed up to 60 months
Overall Survival | From date of CTX130 until date of death due to any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Keegan, PhD, Study Director — CRISPR Therapeutics
Locations (10):
- United States (8):
  - Research Site 2, Duarte, California
  - Research Site 5, Stanford, California
  - Research Site 10, New Haven, Connecticut
  - Research Site 4, Miami, Florida
  - Research Site 9, New York, New York
  - Research Site 8, The Bronx, New York
  - Research Site 1, Houston, Texas
  - Research Site 6, Salt Lake City, Utah
- Research Site 3, Sydney, New South Wales, Australia
- Research Site 7, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iyer SP, Sica RA, Ho PJ, Prica A, Zain J, Foss FM, Hu B, Beitinjaneh A, Weng WK, Kim YH, Khodadoust MS, Huen AO, Williams LM, Ma A, Huang E, Ganpule A, Nagar SD, Sripakdeevong P, Cullingford EL, Karnik S, Dequeant ML, Patel JN, He XS, Li Z, He QA, Mendonez JH, Keegan A, Horwitz SM. Safety and activity of CTX130, a CD70-targeted allogeneic CRISPR-Cas9-engineered CAR T-cell therapy, in patients with relapsed or refractory T-cell malignancies (COBALT-LYM): a single-arm, open-label, phase 1, dose-escalation study. Lancet Oncol. 2025 Jan;26(1):110-122. doi: 10.1016/S1470-2045(24)00508-4. Epub 2024 Nov 29. PMID 39617017
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350